CLINICAL TRIAL: NCT02266823
Title: Program to Improve Care in Complex Chronic Disease
Brief Title: Diabetes CKD Lifestyle Technology Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 14-00563
Record Dates: First submitted 2014-09-18; First posted 2014-10-17 (Estimated); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Chronic Kidney Disease; Diabetes; Obesity
MeSH Terms: conditions — Renal Insufficiency, Chronic; Diabetes Mellitus; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention: Lifestyle A. (Active Comparator): Lifestyle A will receive an iPad loaded with a self-monitoring program used to support vigilance, reduce the information processing requirements, make readily available the information required to make good self-management decisions, provide real-time feedback, and permit targeted counseling in the context within which lifestyle behaviors occur.
  Using Social Cognitive Theory, the study dietitian will counsel participants via videoconferencing software on the iPad. Using the detailed nutritional and physical activity feedback from the self monitoring programs, the dietitian will use SCT to engage the participants in order to initiate healthy behavior change whilst reducing the demands of commuting for in person nutritional counseling.
  Interventions: Behavioral: Social Cognitive Theory
- Intervention: Lifestyle B. (Other): Participants randomized to this group will receive 6 months of routine care followed by a delayed intervention. Lifestyle B will employ the same diet and physical activity prescription as Lifestyle A as described above.
  Using Social Cognitive Theory, the study dietitian will counsel participants via videoconferencing software on the iPad. Using the detailed nutritional and physical activity feedback from the self monitoring programs, the dietitian will use SCT to engage the participants in order to initiate healthy behavior change whilst reducing the demands of commuting for in person nutritional counseling.
  Interventions: Behavioral: Social Cognitive Theory

INTERVENTIONS:
Behavioral: Social Cognitive Theory — The intervention, which combines behavioral counseling with mobile self-monitoring, will be based on SCT which focuses on the role played by self-referent thought in the maintenance of behavior change. Within SCT, behavior change and maintenance are influenced strongly by the individual's perceived self-efficacy.
  Other Names: SCT

SUMMARY:
The purpose of this study is to pilot test an mHealth technology-supported behavioral intervention designed to engage patients with diabetes and concurrent chronic kidney disease (CKD) in multiple behaviors which aim to reduce CKD progression. Participants will be randomized to the 6-month lifestyle intervention or to a wait-list control. The lifestyle intervention will be modeled after that used in the Diabetes Prevention Program (DPP) and the counseling intervention will be based on SCT, which will be paired with mobile technology-based dietary and physical activity monitoring. The wait-list control will receive 6 months of standard medical care followed by a delayed, but less intensive, 6-month intervention.

DETAILED DESCRIPTION:
The purpose of this study is to develop and pilot test a lifestyle intervention in obese individuals with t2dm and concurrent stage 2-4 ckd. The counseling intervention will be based on social cognitive theory and supported by mobile (ipad) self-monitoring. Mobile self-monitoring is featured in the intervention to encourage vigilance to the diet in a manner that is not burdensome, enhance self-efficacy by integrating complex information regarding the ckd dietary regimen with a calorie-restricted diet, and permit real-time monitoring of weight, blood glucose, blood pressure, and self-reported diet and physical activity by the study team.

Specifically, the investigators will develop the methods for and pilot test the ckd lifestyle intervention in stage 2-4 ckd patients and explore the impact of the intervention on: (a) weight and fat mass, (b) blood pressure, (c) physical activity, (d) urinary sodium excretion, (e) serum phosphorus and calcium-phosphorus product, (f) kidney function as measured by serum cystatin-c, and (g) serum lipids. Additionally, we will evaluate the feasibility and acceptability of this intervention in terms of: (h) recruitment and retention, (i) time and cost associated with training ckd patients in technology-based self-monitoring and in delivering the intervention, (j) patterns of self-monitoring adherence over time, and (k) participant satisfaction with the intervention. Finally, we will describe: (l) the extent to which the intervention differentially adversely affects the nutritional health of participants as evidenced by low serum albumin or serum prealbumin; a body mass index (bmi) that falls below 20kg/m2; and subjective assessment of nutritional risk (e.g. Nausea, diarrhea, anorexia).

ELIGIBILITY:
Inclusion Criteria:

* In order to be eligible for the study, the individual must be 40 years of age or older; have a DRG Code of T2DM, GFR of 15-89 ml/min/1.73m2 and a BMI >30 kg/m2. The participant's physician of record will have verified that his/her patient can safely participant in an intervention study that involves weight loss and a goal of 150 minutes/week of moderate physical activity (comparable to brisk walking).

Exclusion Criteria:

* Those with the following characteristics will be excluded by the investigators:

  1. unable or unwilling to provide informed consent; (2) unable to participate meaningfully in an intervention that involves group sessions (e.g., due to uncorrected hearing impairment, non-English-speaking); (3) unable to read or otherwise use an iPad to monitor dietary intake, physical activity, and weight (e.g., blind, illiterate); (4) unwilling to accept randomization assignment; (5) pregnant, or plans to become pregnant in the next 12 months, less than 3 months postpartum, or nursing or within 6 weeks of having completed nursing; (6) weight loss of > 10% in the past 6 months except for postpartum weight loss; and (7) individuals who are institutionalized (e.g., in a nursing home or personal care facility, or those who are incarcerated and have no control over their diet).

will exclude from the study those with underlying diseases which would increase the risk of participating in an intervention involving caloric restriction and physical activity. Such individuals would include those requiring treatment for cancer, exclusive of skin cancer other than melanoma, in the past 2 years; infectious diseases including untreated AIDS and active tuberculosis; uncontrolled hypertension of >190 mmHg SBP or >105 mmHg DBP despite treatment; stroke or TIA in the past 6 months; conditions requiring the use of home oxygen; or other chronic disease or condition likely to limit life span to < 1 year. A recent Institute of Medicine report suggests that reducing dietary sodium below 1,840 mg/day in those with mid- to late-stage heart failure may increase adverse events or mortality. Thus investigators will exclude those with heart failure.

Because of the dietary requirements of a pregnant woman, and the nature of weight loss and gain with pregnancy, inclusion of pregnant women in the study would confound the study results. Those who become pregnant during the study will be withdrawn from the study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2015-10; Primary Completion 2019-11-08 (Actual); Study Completion 2019-11-08 (Actual)

PRIMARY OUTCOMES:
Primary outcome: Weight. Weight will be obtained using a single, calibrated scale. | Change from baseline in weight at 6 months
Primary outcome: Urinary sodium. We will estimate dietary sodium intake from a spot urine sample. | Change from baseline in Urinary sodium at 6 months
Primary outcome: Blood pressure. BP will be obtained using a mercury sphygmomanometer | Change from baseline in Blood pressure at 6 months
Primary outcome: Physical activity. Energy expenditures and minutes devoted to physical activity will be recorded using a FitBit. | Change from baseline in Physical activity at 6 months
Primary outcome: Serum Cystatin-C. Cystatin-C is a serum protein that is used as a biomarker of kidney function | Change from baseline in Cystatin-C at 6 months
Primary outcome: Lipoproteins. We will evaluate the impact of the intervention on serum lipids obtained after a 12-hour fast | Change from baseline in Lipoproteins at 6 months
Primary outcome: Serum Phosphorus and corrected Calcium-Phosphorus product (CaxPO4) will be evaluated from a venipuncture sample. | Change from baseline in Serum Phosphorus and corrected Calcium-Phosphorus product at 6 months
  Corrected CaxPO4 is a measure of metastatic calcification, adjusted for the participant's nutritional status (serum albumin). When serum albumin is < 4 g/dL, the algorithm for corrected CaxPO4 is [Ca + 0.8(4 - serum albumin)]x PO4. When serum albumin if > 4 g/dL, corrected CaxPO4 = CaxPO4. CaxPO4 is obtained with routine monthly labs on all HD patients
Primary outcome: Serum Phosphorus and corrected Calcium-Phosphorus product (CaxPO4) will be evaluated from a venipuncture sample. | Change from baseline in Serum Phosphorus and corrected Calcium-Phosphorus product at 12 months
  Corrected CaxPO4 is a measure of metastatic calcification, adjusted for the participant's nutritional status (serum albumin). When serum albumin is < 4 g/dL, the algorithm for corrected CaxPO4 is [Ca + 0.8(4 - serum albumin)]x PO4. When serum albumin if > 4 g/dL, corrected CaxPO4 = CaxPO4. CaxPO4 is obtained with routine monthly labs on all HD patients
Primary outcome: Weight. Weight will be obtained using a single, calibrated scale. | Change from baseline in weight at 12 months
Primary outcome: Urinary sodium. We will estimate dietary sodium intake from a spot urine sample. | Change from baseline in Urinary sodium at 12 months
Primary outcome: Blood pressure. BP will be obtained using a mercury sphygmomanometer | Change from baseline in Blood pressure at 12 months
Primary outcome: Physical activity. Energy expenditures and minutes devoted to physical activity will be recorded using a FitBit. | Change from baseline in Physical activity at 12 months
Primary outcome: Serum Cystatin-C. Cystatin-C is a serum protein that is used as a biomarker of kidney function | Change from baseline in Cystatin-C at 12 months
Primary outcome: Lipoproteins. We will evaluate the impact of the intervention on serum lipids obtained after a 12-hour fast | Change from baseline in Lipoproteins at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Mary Ann Sevick, ScD, RN, Principal Investigator — NYU School of Medicine
Locations (1):
- NYU Langone Medical Center, New York, New York, United States